CLINICAL TRIAL: NCT00594789
Title: Closing The Post Fracture Care Gap In Manitoba
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Manitoba Patient Access Network Steering Committee (Unknown); The Manitoba Bone Density Program Committee (Unknown)
Responsible Party: Principal Investigator, William D. Leslie, Professor of Medicine and Radiology, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H2007:165
Record Dates: First submitted 2008-01-03; First posted 2008-01-16 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Fractures; Bone densitometry; Dual-energy x-ray absorptiometry
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (physician-only) (Experimental): Physician(s) connected with a fracture that meets study inclusion criteria.
  Interventions: Other: Information letters
- 2 (physician/patient) (Experimental): Physician(s) and patient connected with a fracture that meets study inclusion criteria.
  Interventions: Other: Information letters
- Control (No Intervention): Usual care.

INTERVENTIONS:
Other: Information letters — Information letters under Manitoba Health letterhead will be sent out to physician(s) and/or patient connected with a fracture that meets specific criteria. To address concerns over discontinuous care of patient seen at the time of fracture and for subsequent follow-up, the physician notification will specifically target the individual involved in the initial report to Manitoba Health as well as the primary care physician (using an algorithm developed by the Manitoba Centre for Health Policy). The notification will provide a general recommendation for osteoporosis assessment in addition to a copy of the BMD testing requisition since BMD testing is usually justified in this setting. The notification will not dictate what testing or treatment needs to be performed.
  Arms: 1 (physician-only); 2 (physician/patient)

SUMMARY:
The objective of this study is to evaluate a post-fracture intervention for improving osteoporosis care in older men and women who have suffered a fracture that may indicate the presence of osteoporosis. Although osteoporosis can be identified with a bone mineral density (BMD) test, most individuals with osteoporosis are not diagnosed until they fracture. Post-fracture care often "falls between the cracks" when there is a breakdown in communication between hospital and community, or between specialists and primary care physicians. Often physicians and patients fail to make the connection between an acute fracture and osteoporosis, or the value of secondary prevention strategies. If untreated, there is an extremely high rate of additional fractures after a first osteoporotic fracture. It follows that improving BMD testing and/or treatment in appropriately identified individuals is a necessary step in optimizing post-fracture patient care. Over the next three years we will be testing and optimizing a notification procedure to physicians and/or patients relying upon fracture events reported to the provincial health service (Manitoba Health).

DETAILED DESCRIPTION:
A major 'care gap' exists in the management of patients with fractures suggestive of osteoporosis. Currently, only a small minority of these individuals who are at high risk for recurrent fractures undergo evaluation for possible treatment. We propose to test and optimize a novel approach to address this question, relying upon fracture events reported to provincial health service (Manitoba Health) as a mechanism for osteoporosis case identification and enhancing post fracture care.

Phase 1 (one year duration): individuals meeting the fracture case definition will be randomized to usual care (no intervention), physician notification and physician/patient notification. The notification will provide a general recommendation for osteoporosis assessment. The use of appropriate post-fracture investigations and treatment will be prospectively evaluated.

Phase 2 (up to two years duration): the intervention will be refined and iteratively trialed for all individuals meeting the fracture case definition.

Phase 3: a recommendation for long term maintenance of the post-fracture intervention will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Women and men age 50 and older with one of the following fracture definitions:

  * Hip fracture (physician ICD-9-CM 820-821 plus a procedure code for site-specific fracture reduction or fixation, open or closed)
  * Spine fracture (physician ICD-9-CM code 805), or
  * Humerus fracture (physician ICD-9-CM code 812), or
  * Colles' fracture (physician ICD-9-CM code 813 plus a physician claim for site-specific fracture reduction or fixation, open or closed, or cast application).

Exclusion Criteria:

* Age less than 50.
* Non-Manitoba residents, cancelled Manitoba Health coverage, death or discharge to a personal care home.
* A fracture event in the previous 12 months meeting the study case definition (i.e., only a single notification per year is planned).
* Hip or wrist fractures without a procedure tariff.
* Current treatment with an osteoporosis medication.
* BMD testing within the preceding 3 years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4264 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rates of BMD testing and/or osteoporosis pharmacotherapy in the year post-fracture using the population-based provincial administrative health data repository. | 3 years (Phase 1 analysis at 1 year)

SECONDARY OUTCOMES:
For individuals referred for BMD testing, an evaluation of treatment appropriateness will be performed based upon BMD results and 10-year fracture risk methods. | 3 years (Phase 1 analysis at 1 year)
Repeat fracture rates will be also studied as a secondary endpoint. | 3 years (Phase 1 analysis at 1 year)
An evaluation of post-fracture BMD testing and treatment rates in the years prior to the Phase 1 will also be performed to document practice patterns before the intervention. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William D Leslie, MD MSc, Principal Investigator — Faculty of Medicine, University of Manitoba
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Leslie WD, Metge C. Establishing a regional bone density program: lessons from the Manitoba experience. J Clin Densitom. 2003 Fall;6(3):275-82. doi: 10.1385/jcd:6:3:275. PMID 14514998
- [Background] Caetano PA, Labine L, Klassen P, Dreilich D, Leslie WD. Closing the postfracture care gap using administrative health databases: design and implementation of a randomized controlled trial. J Clin Densitom. 2011 Oct-Dec;14(4):422-7. doi: 10.1016/j.jocd.2011.04.008. Epub 2011 Jul 1. PMID 21723766
- [Background] Leslie WD, LaBine L, Klassen P, Dreilich D, Caetano PA. Closing the gap in postfracture care at the population level: a randomized controlled trial. CMAJ. 2012 Feb 21;184(3):290-6. doi: 10.1503/cmaj.111158. Epub 2011 Dec 19. PMID 22184366
- [Background] Majumdar SR, Lier DA, Leslie WD. Cost-effectiveness of two inexpensive postfracture osteoporosis interventions: results of a randomized trial. J Clin Endocrinol Metab. 2013 May;98(5):1991-2000. doi: 10.1210/jc.2013-1034. Epub 2013 Apr 17. PMID 23596140
- [Derived] Cui Y, Lix LM, Yang S, Morin SN, Leslie WD. A population-based study of postfracture care in Manitoba, Canada 2000/2001-2014/2015. Osteoporos Int. 2019 Oct;30(10):2119-2127. doi: 10.1007/s00198-019-05074-8. Epub 2019 Jul 2. PMID 31267162
- See also: Manitoba BMD Program — http://www.gov.mb.ca/health/primarycare/providers/chronicdisease/bonedensity/index.html